CLINICAL TRIAL: NCT07022028
Title: Ventilator Weaning Practices in Patients Intubated for Guillain-Barré Syndrome or Myasthenia Gravis
Acronym: GUIMAUVE
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GUIMAUVE study
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Myasthenia Gravis; Guillain-Barre Syndrome
Keywords: Myasthenia Gravis; Guillain-Barre syndrome; Ventilator Weaning; Airway Extubation; Intensive Care Unit
MeSH Terms: conditions — Myasthenia Gravis; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients mechanically ventilated for Guillain-Barré syndrome or for myasthenia gravis (two groups)

SUMMARY:
Guillain-Barré syndrome and myasthenia gravis are two neuromuscular diseases that are commonly managed in ICUs that may require different weaning protocols. To date, no study has compared weaning modalities from mechanical ventilation in patients with these two diseases. Our objective was to assess and compare for ventilator weaning modalities between patients mechanically ventilated for Guillain-Barré syndrome or for myasthenia gravis in a large-scale multicenter study.

ELIGIBILITY:
Inclusion Criteria: All patients mechanically ventilated for at least 48 hours for Guillain-Barré syndrome or myasthenia gravis -

Exclusion Criteria: Patients mechanically ventilated less than 48h or intubated for another reason than the neuromuscular disease.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients intubated and mechanically ventilated in ICUs for Guillain-Barré syndrome or myasthenia gravis
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with prolonged weaning | 7 days after the initial separation attempt from the ventilator
  Prolonged weaning defined as still being under mechanical ventilation at least 7 days after the initial separation attempt from the ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud W THILLE, MD, PhD, Principal Investigator — University Hospital of Poitiers
Locations (1):
- CHU de POITIERS, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided